CLINICAL TRIAL: NCT00737854
Title: Free Soft Tissue Graft in Treatment of Oral Lichen Planus
Acronym: TOLP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Qazvin University Of Medical Sciences, Qazvin University Of Medical Sciences . Deputy of Research
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ACTG022
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-08

CONDITIONS: Oral Lichen Planus
Keywords: OLP; Free Soft Tissue Graft; Treatment
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 ARM (Experimental): Otherwise healthy patients with oral lichen planus (precancerous/erosive OLP)
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Procedure: Surgical resection — 20 patients with OLP will be selected for this study. Before this routine treatment modalities had been attempted. Removal of possible triggering drug was also considered. Local ethical committee approval will be obtained before the trial starts. Surgical procedure includes: removal of the tissue up to submucosa (containing antigenic properties that caused OLP). A specimen will be sent for histopathologic analysis. The graft sliced from healthy mucosa also up to submucosa. Then the graft trimmed on a gauze soaked in saline and adapted to recipient site. The graft was sutured in position. Checking will be done after 1 week and every two months up to 1 year. Punch biopsy will be done in 1 year after surgery for histopathologic investigations.
  Other Names: surgical resection of OLP

SUMMARY:
Oral lichen planus is a common chronic mucocutaneous disease with various clinical forms. Erosive-ulcerative forms usually cause symptoms of pain and discomfort. The most important complication of OLP is development of oral squamous cell carcinoma, although this is a very controversial matter. various treatments have been suggested for OLP but their results are unsatisfactory. Through the experiences of the investigators, corticosteroids (in any form)is not a wise option for treating OLP and has many side effects . More over, immunosuppressive therapy did not influence the risk for oral cancer. The purpose of the study is to determine the efficacy of free soft tissue graft in the treatment of precancerous and symptomatic lesions of OLP. Removal of the lesions up to submucosa has been done. The graft sliced from healthy mucosa also up to submucosa. Then graft will be sutured in position.

According to other authors, basal epithelial layers of the graft remain intact and represent the focus of re-epithelization. New epithelial cells migrate over the basal membrane and appear to guide it by proliferation, will generate new epithelium. The wound is re-epithelialized by proliferation of surrounding healthy epithelial cell, therefore, not contaminated by modified antigens of the cell membrane that are theoretically responsible for lymphocyte aggression. The healthy graft remains free of lesions and appears clinically healthy.

DETAILED DESCRIPTION:
Oral lesions in OLP are chronic ,rarely undergo spontaneous remission, are potentially premalignant and are often a source of morbidity. recent study does not support that non reticular OLP are more predisposed to malignant change. Moreover , immunosuppressive therapy did not influence the risk for oral cancer. in general ,all treatment should be aimed at eliminating precancerous lesions ,alleviating symptoms ,and potentially decreasing the risk of malignant transformation. Although the cause of OLP is unknown , it is generally considered to be an immunologically mediated process that microscopically resembles a hypersensitivity reaction .it is characterized by an intense T cell infiltrate localized to epithelium-connective tissue interface. the purpose of the study is to determined the efficacy of free soft tissue graft in treatment of precancerous and symptomatic lesions of OLP. so removal of the lesions up to submucosa will be done. the graft sliced from healthy mucosa also up to submucosa . then graft will be sutured in position.

According to other authors, basal epithelial layers of the graft remain intact and represent the focus of reepithelialization. new epithelial cell migrate over the basal membrane and appear to guide it and by proliferation ,will generate new epithelium. so the wound is re-epithelialized by proliferation of surrounding healthy epithelial cell, therefore, not contaminated by modified antigens of the cell membrane that are theoretically responsible for lymphocyte aggression so the healthy graft remains free of lesions and appears clinically healthy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed symptomatic oral lichen planus: WHO histological criteria in combination with clinical appearance will be used for diagnosis
* Previous routine treatment modalities has been attempted including steroids and immunomodulatory or antioxidant agents. i.e patients who had resistant lesions to routine treatment .removal of possible triggering drugs was also considered.
* Patients of both sexes between 40 to 70 year's old
* Patients who have symptoms such as burning sensation, pain
* Patients who have localized precancerous lesions such as atrophic-erosive/plaque like lichen planus with diameter lesser than 2 cm
* Patients who agree to this treatment
* Patients who are willing for evaluation in first week after surgery and every two month for 1 years
* Patients who agree to final punch biopsy for histopathologic evaluation

Exclusion criteria:

* Patients who unable to undergo oral surgery
* Patients suffering from any localized or systemic disease
* Pregnant patients
* Smokers
* Patients who can not continue the study for private or social reasons
* Patients with generalized oral lichen planus

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Relief of sign & symptoms (every 2 month up to 1 years) | 1 year

SECONDARY OUTCOMES:
Relief of sign & symptoms and no positive histopathologic features of OLP | (time frame 1 years)

CONTACTS AND LOCATIONS:
Overall Officials: Farshid Rayati, DDS, Study Director — Qazvin University Of Medical Sciences; Tuba(Aida) Karagah, DDS, Principal Investigator — QUMS; Farshid Rayati, DDS, Study Chair — QUMS; Saeid Asefzadeh, PHD, Study Chair — QUMS; Poopak masumi, DDS-MS, Study Director — QUMS; pourya falah, student, Principal Investigator — QUMS
Locations (1):
- Qazvin University of Medical Sciences, Qazvin, Qazvin State, Iran